CLINICAL TRIAL: NCT04952363
Title: The Effect of Whole Body Vibration Training on Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Whole-body Vibration on Mucus Clearance, the Quality of Life, and Exercise Capacity for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-E(Ⅱ)-20170267
Record Dates: First submitted 2021-06-24; First posted 2021-07-07 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HFCWO+WBVT (Experimental): Subjects received HFCWO+WBVT intervention twice a week for a period of 8 weeks
  Interventions: Device: A vertical vibration platform PowerVibe Zen Pro 5900; Device: HFCWO
- HFCWO only (Active Comparator): Subjects received HFCWO intervention twice a week for a period of 8 weeks
  Interventions: Device: HFCWO

INTERVENTIONS:
Device: A vertical vibration platform PowerVibe Zen Pro 5900 — Subjects received the interventions twice a week for 8 weeks. HFCWO+WBVT group received additional 30 minutes WBVT treatment. In every WBVT session, three rounds of 3 minutes of vibration (amplitude: 2 mm; frequency: 20 Hz) were provided, with a 60-second rest between rounds.
  Arms: HFCWO+WBVT
Device: HFCWO — Subjects received the interventions twice a week for 8 weeks. The HFCWO was delivered by a respiratory therapist using a percussive vest at 10-13 Hz oscillating frequency and at a pressure setting of 2 cm H2O. The treatment duration was 25 minutes, and the participants remained in a sitting position.

SUMMARY:
Although whole body vibration (WBV) is mainly designed to promote neuromuscular function, however, because of its vibration characteristics, whether it can provide additional effects on the sputum clearance for chronic obstructive pulmonary (COPD) disease patients, thereby improving the quality of life, and exercise capacity is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD at the outpatient thoracic medicine clinic
* Need HFCWO as judged by the doctor

Exclusion Criteria:

* Acute COPD exacerbation within the previous 4 weeks,
* Contraindication for WBVT (e.g., artificial joint replacement, a history of deep vein thrombosis, or known aortic aneurysm)
* Inability to perform squatting exercises
* Acute disc disease
* Inability to complete the 6MWT

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
FVC | 8 weeks
  forced vital capacity tested in pulmonary function test (Liters)
FEV1 | 8 weeks
  forced expiratory volume in 1 second in pulmonary function test (Liters)
FEV1/FVC | 8 weeks
  forced expiratory volume in 1 second divided by forced vital capacity in pulmonary function test (%)
FVC(% pred) | 8 weeks
  percentage of predicted FVC value (% pred)
FEV1(% pred) | 8 weeks
  percentage of predicted FEV1 value (% pred)
6 min walk distance | 8 weeks
  the distance walked in 6 minutes (m)
Predicted distance | 8 weeks
  percentage of the predicted 6 minute walk test distance (%pred)
Distance-Saturation Product (DSP) | 8 weeks
  the product of distance walked and lowest oxygen saturation during the 6-min walk test (m%)
1 min STST | 8 weeks
  the number of repetitions performed in the 1-min sit-to-stand test (rep.)
5-rep STST | 8 weeks
  the complete time for the 5-repetition sit-to-stand test (sec)
Muscle strength test1 | 8 weeks
  Maximal force output for biceps femoris muscle (lbs)
Muscle strength test2 | 8 weeks
  maximal force output for quadriceps muscle (lbs)
Sputum self-assessment scale | 8 weeks
  questionnaire of sputum volume, it contained three items (0-25 mL/d, 25-50 mL/d, and 50-100 mL/d) as a checklist
X-ray score | 8 weeks
  the evaluation of the chest radiography based on the sputum impaction score, scores ranging from 0 to 18. A decrease in score represented an improvement in sputum in each area.
modified Medical Research Council (mMRC) | 8 weeks
  questionnaire of dyspnea, scores ranging from 0 (low degree of dyspnea) to 4 (high degree of dyspnea)
chronic obstructive pulmonary disease assessment test (CAT) | 8 weeks
  questionnaire of COPD symptoms, scores ranging from 0 to 40, higher scores indicating more severe impact of COPD on their life
Saint George Respiratory Questionnaire (SGRQ) | 8 weeks
  questionnaire of overall health, daily life, and perceived well-being, scores ranging from 0 (no health impairment) to 100 (maximum health impairment)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan